CLINICAL TRIAL: NCT07054658
Title: Evaluation of Allogenic Bone Ring Graft With Simultaneous Implant Placement for Vertical Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ibrahim Taha Hussein, Principal Investigator, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD-3-24-2166
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Posterior Mandible With Deficient Ridge Height
Keywords: vertical ridge augmentation; bone ring technique

STUDY DESIGN:
Intervention Model Description: Participants in this study received an allogenic bone ring graft for vertical ridge augmentation, with simultaneous dental implant placement
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogenic Bone Ring With Simultaneous Implant Placemen (Experimental): Patients received vertical ridge augmentation using a customized allogenic bone ring graft with simultaneous dental implant placement in the posterior mandible
  Interventions: Procedure: Allogenic Bone Ring Graft With Simultaneous Implant Placement

INTERVENTIONS:
Procedure: Allogenic Bone Ring Graft With Simultaneous Implant Placement — A surgical procedure involving vertical ridge augmentation using an allogenic bone ring combined with simultaneous dental implant placement in the posterior mandible. The technique allows one-stage treatment of vertical bone defects without the need for autogenous bone harvesting.

SUMMARY:
This clinical trial aimed to evaluate the effectiveness of vertical ridge augmentation using customized allogenic bone ring grafts with simultaneous dental implant placement in the posterior mandible. The procedure is designed to address vertical bone deficiencies without the need for autogenous bone harvesting, thereby reducing patient morbidity and surgical complexity. The study assessed clinical outcomes including bone gain, implant stability, and over a 6-month period and inflammation, infection, pain and neurosensory changes where assessed for 4 weeks.

DETAILED DESCRIPTION:
This study investigated the clinical outcomes of vertical ridge augmentation using allogenic bone rings in combination with simultaneous implant placement for the treatment of posterior mandibular bone defects. Traditional ridge augmentation techniques often require two-stage surgeries and autogenous bone harvesting, which may increase patient morbidity and prolong healing. In contrast, the allogenic bone ring technique provides a one-stage approach by allowing vertical augmentation and implant placement to be performed simultaneously.

The study was designed as a prospective, single-arm clinical trial. Eligible patients aged 18 years or older, presenting with vertical bone deficiencies in the posterior mandible, were recruited from the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Tanta University. The primary outcome was vertical bone gain measured radiographically at 6 months postoperatively. Secondary outcomes included implant stability (measured by IST), soft tissue healing, and postoperative complications. Patients were followed clinically and radiographically to evaluate the success of the grafting procedure and implant integration.

ELIGIBILITY:
Inclusion Criteria:

* Participants with vertical alveolar ridge atrophy in the posterior mandible who are motivated, cooperative, and have good oral hygiene.
* Minimum of 7 mm remaining bone height from the crest of the alveolar ridge to the inferior alveolar canal.
* Patients with adequate remaining interarch space

Exclusion Criteria:

* Prior local radiation therapy.
* Soft and hard tissue pathology at the operation site.
* Systemic diseases that might affect bone healing and osseointegration (e.g., uncontrolled diabetes)..
* smokers who consume 20 or more cigarettes per day.
* patients on anti-resorptive drugs (eg: bisphosphonates and denosumab).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Vertical Bone Gain in mm | 6 months postoperatively
  The vertical bone gain was measured radiographically using CBCT imaging to evaluate the effectiveness of the allogenic bone ring graft in augmenting vertical bone height in the posterior mandible

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim T Hussein, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Rafic R Beder, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Khaled A Saad, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Maram N Breshah, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Derived] Hussein IT, Beder RR, Saad KA, Breshah MN. Evaluation of allogenic bone ring graft with simultaneous implant placement for vertical ridge augmentation. Oral Maxillofac Surg. 2025 Dec 1;30(1):4. doi: 10.1007/s10006-025-01487-4. PMID 41320709